CLINICAL TRIAL: NCT05053958
Title: Patients' Satisfaction and Aesthetic Outcomes of Single Implant Restorations in Aesthetic Zone Using Superimposition of Intra-Oral Scan and CBCT.
Brief Title: Using Superimposition of Intra-Oral Scan and CBCT in Single Implant Restorations in Aesthetic Zone.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Dina Mohamed Aboulftouh Ahmed, assistant lecturer of fixed prosthodontics department, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: P-CR-21-06
Record Dates: First submitted 2021-09-08; First posted 2021-09-23 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Dental Implant; Patient Satisfaction
Keywords: digital Implantology; patient reported outcomes; guided surgery; aesthetic outcomes; accuracy
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implant planning without using superimposition of intraoral scan and CBCT. (No Intervention): Patients will receive a pre-operative CBCT examination. Implants will be inserted using freehand drilling protocol. The implants will be placed using flapless technique with the reference of neighboring teeth and 3D radiographic information.
- Implant planning using superimposition of intraoral scan and CBCT. (Active Comparator): Patients will receive a pre-operative CBCT examination and optical scan of the oral tissues by intra-oral scanner. Digital Imaging and Communications in Medicine (DICOM) file from the CBCT examination and the Standard Tessellation Language (STL) file from the optical scan will be imported and merged in implant planning software. The virtual implant planning will be performed. The surgical guide and prosthesis are designed according to the virtual plan.
  Interventions: Other: superimposition of DICOM file from CBCT and STL file of Intraoral scanner

INTERVENTIONS:
Other: superimposition of DICOM file from CBCT and STL file of Intraoral scanner — These files will be imported in implant planning software,and virtual implant planning will be performed.
  Arms: Implant planning using superimposition of intraoral scan and CBCT.

SUMMARY:
This study will be performed to evaluate patients'satisfaction and aesthetic outcomes of single implant restorations in aesthetic zone by using superimposition of intra-oral scan and CBCT.

DETAILED DESCRIPTION:
The accurate transfer of an ideal implant position from virtual planning to the actual implant site is essential for protecting vital structures as well as optimizing esthetic and functional outcomes.With the introduction of 3D imaging and implant planning software, preoperative design for a "prosthesis-driven" implant position becomes a reality.

The initial stage is digital image acquisition, which can be from extra-oral means such as cone beam computed tomography (CBCT) and laboratory scanners, or intraoral means such as intraoral scanners.

Image fusion or superimposition of the STL data obtained from the optical scanning, with the DICOM data obtained from the CBCT, is performed by matching the common reference points prior to implant planning.

The superimposed images enable virtual implant planning, while taking the surrounding anatomic structures and future prosthetic needs into consideration.

To conduct the present study, the following will be used:

1. DICOM file of CBCT for examination of single implant in aesthetic zone.
2. STL file of optical scanning for examination of single implant in aesthetic zone.
3. An implant planning software.
4. One type of dental implant.

ELIGIBILITY:
Inclusion Criteria:

1. At least 1 tooth having missed within 3-4 months or to be extracted in anterior zone, and the remaining teeth are adequate to support the surgical template.
2. Sufficient bone tissue to insert an implant without any need for augmentation (the residual bone height ≥ 10 mm, the buccolingual width ≥ 7 mm, and the labial bone plate is complete without bone dehiscence and fenestration).
3. Good treatment compliance.

Exclusion Criteria:

1. Presence of uncontrolled systemic diseases, infection, or inflammation around the implant sites.
2. Pregnancy or lactation.
3. Poor oral hygiene habits.
4. Psychiatric problems, alcohol, tobacco (>10 cigarettes per day) or drug abuse.
5. Severe bruxism or clenching.
6. Not able to complete the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score | 0-3 month
  A total of seven variables (mesial papilla, distal papilla, level of soft-tissue margin, soft-tissue contour,alveolar process deficiency, soft-tissue color,and soft-tissue texture) assessing soft tissue around single implant supported restoration with a score of 0 to 2 (0 representing the poorest and 2 the best result) . The maximum score of 14 points reflects perfect implant esthetics with that of the contra lateral tooth.
Implant Crown Aesthetic Index | 0-3months
  A total of nine variables ( Width ,Length ,Labial convexity ,Color/translucency,Surface,Labial margin ,Papillae, Contour of the labial surface,Color and surface) assessing implant crown and soft tissue esthetics using the score of 0=no deviation, 1= small deviation and 5=large deviation. The maximum score of 45 points reflects perfect implant esthetics with that of contra lateral and adjacent tooth.
White Esthetic Score | 0-3 months
  A total of five variables (tooth form,tooth volume/outline, color, surface texture and translucency) assessing implant crown esthetics using a score from 0 = worst to 2 = best result. The highest possible score of 0 reflects perfect implant esthetics with that of the contra-lateral tooth.
Peri-Implant and Crown Index (PICI) | 0-3months
  A total of six variables (Papillae ,Zenith ,Root convexity o f the peri implant mucosa and Shape ,Color ,Characterization of the implant crown )assessing crown,mucosa and Overall crown and mucosa compared to contra lateral tooth using 100 mm visual analogue scale.
Patient satisfaction level | 3months
  using a subjective outcome questionnaire filled out by patient him/herself

CONTACTS AND LOCATIONS:
Overall Officials: Osama S Abdel Ghani, Study Director — Professor & Head of Crowns and Bridges Department Faculty of Dental Medicine for Girls; Roqaia M Alassar, Study Director — Lecturer of Crowns and Bridges Faculty of Dental Medicine for Girls
Locations (1):
- Al-Azhar University, Cairo, Egypt